CLINICAL TRIAL: NCT01841255
Title: UMOX™: A New Device for Preoxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Louis-Philippe Fortier, Chief of Staff, Anesthesiology Dep., Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06108
Record Dates: First submitted 2013-02-27; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Preoxygenation; Device; Tolerability; Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tidal breathing using the facemask (Sham Comparator): Control
  Interventions: Device: facemask
- Tidal volume breathing with the UMOXTM, device, no instruction (Experimental): First experimental measure
  Interventions: Device: Mouthpiece (Umox)
- Tidal volume breathing with the UMOXTM device, instructions (Experimental): Second experimental measure
  Interventions: Device: Mouthpiece (Umox)
- Tidal volume breathing with the UMOXTM, device, nose clip (Experimental): Third experimental measure
  Interventions: Device: Mouthpiece (Umox)

INTERVENTIONS:
Device: Mouthpiece (Umox) — Device used to perform preoxygenation in the operating room context
  Other Names: Umox
  Arms: Tidal volume breathing with the UMOXTM device, instructions; Tidal volume breathing with the UMOXTM, device, no instruction; Tidal volume breathing with the UMOXTM, device, nose clip
Device: facemask
  Arms: Tidal breathing using the facemask

SUMMARY:
Background - Preoxygenation is performed before general anesthesia to increase the oxygen reserves of the body and prolong the safe period of apnea without hypoxia. However, it is often impossible to obtain a perfect face mask fit, and optimal end-tidal fractional oxygen concentration (EtO2) are not attained. The investigators designed a new oropharyngeal preoxygenation device, UMOX™, to avoid leaks during preoxygenation. In this study, the investigators compared the efficacy of UMOX™ with that of a conventional face mask.

Methods - In 50 healthy volunteers breathing 100% oxygen from a circle absorber system for a 5 minute-period, the investigators compared preoxygenation using the 1) a conventional mask; 2) UMOX™ without any instruction; 3) UMOX™ with instruction on mouth breathing; and 4) UMOX™ with a nose clip, in random order. Each subject underwent all steps with a 10-minute rest period of room air breathing between each step. Inspired and end-tidal respiratory gases were measured every 10 seconds. EtO2 variation was analyzed using Anova.

DETAILED DESCRIPTION:
This study was as a single center, crossover, randomized trial. Following approval from research and ethics committee from our hospital and written consent from healthy subjects recruited, 50 consenting volunteers were enrolled over a three-month period, from: September 29, 2008 to November 5, 2008.

Subjects enrolled were of both genders, smokers and non-smokers, American Society of Anesthesiologists (ASA) physical status I or II, 18 to 65 years old. Nonrecruitment depended on the presence of any craniofacial abnormality, facial hair (beard or moustache) or absence of teeth. Well-controlled non-severe asthma was not a criterion for exclusion.

The trial was conducted in an operating room, using the Dräger Fabius GS (Dräger, Canada), anesthesia machine in a usual set up with the operating table. The investigators used a, patient circuit system consists of 1.5-L lime soda absorber connected to disposable corrugated tubing and a 2-L breathing bag. Gases were analyzed through a Marquette Medical Systems™ SAM module (GE Healthcare), volumes monitored with a GE Respirator Mechanics-M (GE Healthcare) and SpO2 measured with a Nellcor™ (Covidien) pulse oximetry positioned on a finger. Preoxygenation procedures were explained to the subjects and ample time was allowed so they could become familiar with the mask and mouth piece. Set up for the measure was conducted by the same experimenter. Subjects laid supine and preoxygenation was performed with fresh gas flow: 100% oxygen (O2) 10L/minute, administered trough facemask or mouth piece sequentially in a random order. Randomization was established with a random assignment table (ww.randomization.com). The envelope was open as the subject entered the operating room (OR). At the beginning and between each step, the anesthesia circuit was flushed with 100% (O2). Each subject went through all steps in random order, each requiring a 5-min period of: 1) tidal breathing using the facemask (TVFM); 2) tidal volume breathing with the UMOXTM mouthpiece (TVMP); 3) tidal volume breathing with the UMOXTM mouthpiece and verbal instructions to favor mouth breathing (TVMPMB); (4) tidal volume breathing with the UMOXTM mouthpiece and a nose clip (TVMPNC). The experimenter conducting the steps instructed participants to create a seal with their lips around the mouthpiece and readjusted the facemask when the subject signalled a discernable leak. Each step was interrupted by 10 minutes of breathing normal room air to allow for return to original respiratory status. Continuous recording of experimental measures, displayed on the anesthesia monitoring system, was done on digital films (Canon PowershotS5 IS™). For the purpose of our trial, 10 seconds intervals were considered adequate for following preoxygenation trends. End-tidal O2 was measured continuously for 5 min. We have also evaluated the level of satisfaction of the subject with each technique using a 1-4 scale.Participants were asked to asses their comfort by showing the associated number with their fingers. Finally we described the performance of the facemask ventilation technique as reported by the experimenter on a scale of 1 to 4.Primary outcome was the end-tidal O2 at the end of the 5-minutes preoxygenation period. Secondary outcomes included endtidal O2 as a function of time, the number of subjects reaching at least 87% EtO2, subject satisfaction and ease of ventilation.

Based on the few studies available on different preoxygenation technques, the end-tidal oxygen fraction standard deviation can range from 5% to about 20% depending on the device used for preoxygenation3,4,14,15. Assuming a 12% value for standard deviation, sample size calculations were made for Type I and Type II errors of 5% and 20%, respectively (power of 80%). From these numbers and taking account that we would rely on multiple comparisons, the power analysis suggested that 50 subjects would allow us to find a difference between groups around 9%. The 9nvestigators analyzed the EtO2 final value with one-way ANOVA followed by the Tukey's Multiple Comparisons test. Percentage of participants reaching at least 87% EtO2 are described with survival curves compared with Kaplan-Meier log rank test. Tolerance is presented using Kruskal-Wallis with Dunn's Multiple Comparisons test.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* smokers and non-smokers
* American Society of Anesthesiologists (ASA) physical status I or II
* 18 to 65 years old.

Exclusion Criteria:

* Presence of any craniofacial abnormality
* facial hair (beard or moustache) or absence of teeth.
* Well-controlled non-severe asthma was not a criterion for exclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measurement was the evolution of endtidal oxygen fraction during a 5 minute preoxygenation procedure, measurements were done continuously, maximum values were recorded | The four steps were done sequentially, each step consisted of a 5 minute recording period under specific conditions, followed by a 10 minute pause before the next step
  The goal of this study is to compare the efficacy of preoxygenation using the conventional mask with the mouthpiece of the UMOX™ oropharyngeal device. The primary outcome measurement was endtidal oxygen fraction. The investigators also evaluated the respective tolerability of the two preoxygenation instruments in healthy volunteers. The measures were not part of a surgical procedure, participants were volunteers participating in this experimental design. No follow-up step was included in this protocol.

SECONDARY OUTCOMES:
The investigators also evaluated the respective tolerability of the two preoxygenation instruments in healthy volunteers with a short questionnaire | The four steps were done sequentially, each step consisted of a 5 minute recording period under specific conditions, followed by a 10 minute pause before the next step

CONTACTS AND LOCATIONS:
Overall Officials: Louis P Fortier, MD, MSc, Principal Investigator — Université de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada